CLINICAL TRIAL: NCT04849806
Title: Dissecting the Nature and Determinants of Sympathetic Nerve Activity in Patients With COPD
Brief Title: Sympathetic Nerve Activity Predictors in Patients With Chronic Obstructive Pulmonary Disease
Acronym: SNAP-COPD
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: DFG - Deutsche Forschungs Gemeinschaft (German Research Foundation) (Unknown)
Responsible Party: Principal Investigator, Jens Spießhöfer, Jens Spiesshoefer, MD, PhD Candidate, Group head Respiratory Physiology, RWTH Aachen University
Other Study IDs: CTCA 20-423
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COPD; Sympathetic Nervous System Diseases; Catecholamine; Overproduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples based on venous puncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients (n=100): The following parameters will be determined in 100 consecutive patients with COPD without established cardiovascular disease (i.e. without an indication for beta blocker therapy or other pharmacological treatments attacking on the neurohormonal pathways like angiotensin-converting enzyme inhibitors or mineralocorticoid receptor antagonists).
  1. OSA severity.
  2. Determination of PH and right HF severity (defined as tricuspid annular plane systolic excursion ≤14 mm) and pulmonary arterial pressure (PAsys) using transthoracic echocardiography;
  3. Comprehensive lung function and inspiratory muscle function testing ;Assessment of daytime hypoxia (PaO2 <55 mmHg) and hypercapnia (PaCO2 >45 mmHg) using capillary blood gas analysis;
  4. Assessment of systemic inflammation
  Interventions: Diagnostic Test: Assessments of the sympathetic nerve activity axis; Diagnostic Test: OSA severity; Diagnostic Test: Determination of PH and right HF severity; Diagnostic Test: Comprehensive lung function and inspiratory muscle function testing.; Diagnostic Test: Assessment of systemic inflammation
- Controls (n=35): (and in a group of healthy controls [3:1] matched for age, sex and BMI).
  Interventions: Diagnostic Test: Assessments of the sympathetic nerve activity axis; Diagnostic Test: OSA severity; Diagnostic Test: Determination of PH and right HF severity; Diagnostic Test: Comprehensive lung function and inspiratory muscle function testing.; Diagnostic Test: Assessment of systemic inflammation

INTERVENTIONS:
Diagnostic Test: Assessments of the sympathetic nerve activity axis — For assessment sympathovagal balance (SVB), HRV and dBPV will be analysed using a 3-lead electrocardiogram (sampling rate 1000Hz) and a continuous non-invasive arterial blood pressure signal (CNAP® technology, sampling rate 100Hz). HRV (ms2 based on continuously recorded variability in RR intervals) and (diastolic) BPV (expressed as mmHg2 based on continuously recorded variability in diastolic BP) will be computed by time domain analysis and by frequency domain analysis and presented as the high frequency component (HF; 0.15-0.4 Hz), low frequency component (LF; 0.04-0.15 Hz), their relative ratio (LF/HF), and the very low frequency component (VLF; 0.0-0.04 Hz) for both HRV and dBPV .
  Muscle SNA will be recorded via a tungsten microelectrode carefully placed in the peroneal nerve. Plasma catecholamines will also be assessed.
Diagnostic Test: OSA severity — OSA is defined as apnoea-hypopnoea index [AHI] >15/h and obstructive apnoea index [OAI] >5/h) and sleep architecture
Diagnostic Test: Determination of PH and right HF severity — (defined as tricuspid annular plane systolic excursion ≤14 mm) and pulmonary arterial pressure (PAsys) using transthoracic echocardiography
Diagnostic Test: Comprehensive lung function and inspiratory muscle function testing. — Respiratory Muscle strength and function testing as previously established by our group and Assessment of daytime hypoxia (PaO2 <55 mmHg) and hypercapnia (PaCO2 >45 mmHg) using capillary blood gas analysis.
Diagnostic Test: Assessment of systemic inflammation — Based on blood samples taken.

SUMMARY:
The project will be pursued in our respiratory, autonomic nervous system physiology laboratory (Respiratory, autonomic nervous system physiology laboratory, Department of Pneumology and Intensive Care Medicine, RWTH Aachen University Hospital; Head of Department: Professor Michael Dreher).

Overactivity of the sympathetic nerve activity (SNA) axis with "centrally" increased heart rate and peripheral vasoconstriction is a known phenomenon in patients with systolic heart failure (HF) and has recently been described in patients with primary lung disease as seen in chronic obstructive pulmonary disease (COPD).

However, systematic analyses on this clinically relevant topic are currently lacking.

Thus, using a comprehensive, multimodal approach and state-of-the-art technology, this research project is designed to determine the extent and nature of increased SNA in COPD (AIM 1) and evaluate the underlying mechanisms (AIM 2).

The project will address the following hypotheses:

1. In COPD, concomitant obstructive sleep apnea is independently associated with increased SNA.
2. Precapillary pulmonary hypertension (PH), inspiratory muscle dysfunction and systemic inflammation describe a COPD phenotype characterised by increased SNA with a different subtype.

DETAILED DESCRIPTION:
The project will be pursued in our respiratory, autonomic nervous system physiology laboratory (Respiratory, autonomic nervous system physiology laboratory, Department of Pneumology and Intensive Care Medicine, RWTH Aachen University Hospital; Head of Department: Professor Michael Dreher).

Overactivity of the sympathetic nerve activity (SNA) axis is a known phenomenon in patients with systolic heart failure (HF) and has recently been described in patients with primary lung disease as seen in chronic obstructive pulmonary disease (COPD).

Thus, insights into the nature of and factors involved in increased SNA in COPD are urgently needed.

Potentially obstructive sleep apnea (OSA) with not only repetitive obstructions but also additional hypoxia and poor sleep quality additively increase SNA in COPD. In addition, inspiratory muscle dysfunction (if adequately measured by magnetic diaphragm stimulation studies and comprehensive diaphragm ultrasound) with related hypercapnia, pulmonary hypertension (PH) and systemic inflammation all likely also impact on SNA in COPD.

However, systematic analyses on this clinically relevant topic are currently lacking.

Thus, using a comprehensive, multimodal approach and state-of-the-art technology, this research project is designed to determine the extent and nature of increased SNA in COPD (AIM 1) and evaluate the underlying mechanisms (AIM 2). The project will address the following hypotheses:

1. In COPD, concomitant OSA with poor sleep is independently associated with increased SNA,.
2. PH, inspiratory muscle dysfunction and systemic inflammation describe a COPD phenotype characterised by increased SNA, manifesting differently.

To test these hypotheses COPD patients without an established cardiovascular disease will be enrolled and the extent, nature and mechanism of SNA increase compared with healthy controls matched in a 3:1 ratio for age, sex and body mass index (BMI).

Invasive assessment of muscle SNA to the point of single unit recordings with analysis of single postganglionic sympathetic firing, and hence SNA drive to the peripheral vasculature, is the gold standard for quantification of SNA in humans but is only available in a few centres worldwide because it is costly, time consuming and requires a high level of training.

A small substudy will investigate the short term acute treatment effects of non-invasive ventilation and oxygen supplementation on SNA in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Ability and willingness to give informed consent to participate in the study

Exclusion Criteria:

* Atrial fibrillation
* Active pacing of the heart by a cardiac pacemaker (i.e. no intrinsic heart rate)
* Clinically pre-established cardiovascular disease (e.g. arterial hypertension or systolic heart failure)
* In-patient stay in the hospital within the last 4 weeks prior to the study examination date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients (n=60) Controls (n=20) COPD patients without an established cardiovascular disease will be enrolled and the extent, nature and mechanism of SNA increase compared with healthy controls matched in a 3:1 ratio for age, sex and body mass index (BMI).
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessments of the sympathetic nerve activity axis (Non invasive) | 2 years
  sympathovagal balance (SVB), HRV and dBPV will be analysed using a 3-lead electrocardiogram (sampling rate 1000Hz) and a continuous non-invasive arterial blood pressure signal (CNAP® technology, sampling rate 100Hz). HRV (ms2 based on continuously recorded variability in RR intervals) and (diastolic) BPV (expressed as mmHg2 based on continuously recorded variability in diastolic BP) will be computed by time domain analysis and by frequency domain analysis and presented as the high frequency component (HF; 0.15-0.4 Hz), low frequency component (LF; 0.04-0.15 Hz), their relative ratio (LF/HF), and the very low frequency component (VLF; 0.0-0.04 Hz) for both HRV and dBPV .
Assessments of the sympathetic nerve activity axis (Invasive) | 2 years
  Muscle SNA will be recorded via a tungsten microelectrode carefully placed in the peroneal nerve Plasma catecholamines will be assessed Muscle SNA will be recorded via a tungsten microelectrode carefully placed in the peroneal nerve Plasma catecholamines will be assessed Muscle SNA will be recorded via a tungsten microelectrode carefully placed in the peroneal nerve. Plasma catecholamines will be assessed

SECONDARY OUTCOMES:
OSA severity | 2 years
  See above
Determination of PH and right HF severity | 2 years
  See above
Comprehensive lung function and inspiratory muscle function testing as previously described by our group | 2 years
  See above
Assessment of systemic inflammation | 2 years
  See above

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Professor, Study Director — RWTH Aachen University; Jens Spiesshoefer, MD, Principal Investigator — RWTH Aachen University; Binaya Regmi, MD, Study Chair — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spiesshoefer J, Becker S, Tuleta I, Mohr M, Diller GP, Emdin M, Florian AR, Yilmaz A, Boentert M, Giannoni A. Impact of Simulated Hyperventilation and Periodic Breathing on Sympatho-Vagal Balance and Hemodynamics in Patients with and without Heart Failure. Respiration. 2019;98(6):482-494. doi: 10.1159/000502155. Epub 2019 Aug 28. PMID 31461730
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Background] Dreher M, Neuzeret PC, Windisch W, Martens D, Hoheisel G, Groschel A, Woehrle H, Fetsch T, Graml A, Kohnlein T. Prevalence Of Chronic Hypercapnia In Severe Chronic Obstructive Pulmonary Disease: Data From The HOmeVent Registry. Int J Chron Obstruct Pulmon Dis. 2019 Oct 18;14:2377-2384. doi: 10.2147/COPD.S222803. eCollection 2019. PMID 31695357